CLINICAL TRIAL: NCT04264416
Title: Effects of 16 Weeks of Whole-Body Electromyostimulation on Stability, Strength and Golf Performance in Amateur Golfers - A Randomized Controlled Study
Brief Title: Effects of Whole-Body Electromyostimulation on Golf Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMSGOLF
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Golf Specific Performance; Muscle Strength; Trunk Stability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants conducting the assessments and/or analyzed the data are unaware if the status of the participants (WB-EMS vs control) and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-Body Electromyostimulation (Experimental): 16 weeks of dynamic WB-EMS: one supervised session per week, 20 min session; impulse-frequency: 85 Hz; impulse breadth 350 µs; intermittent 4-6 s; of impulse - 4 s of impulse break; impulse intensity RPE 7 (hard+ to very hard) on Borg CR 10 Scale.
  Interventions: Device: WB-EMS
- Non exercising control (No Intervention): ...maintained physical activity and exercise habits during the study period.

INTERVENTIONS:
Device: WB-EMS — 16 weeks of WB-EMS
  Other Names: Whole Body Electromyostimulation
  Arms: Whole-Body Electromyostimulation

SUMMARY:
Golf is becoming increasingly popular in Germany. However, the biomechanical and motor challenge of golf should not be underestimated. Nevertheless, only very few amateur golfers carry out serious preparation and conditioning as part of a strength/stabilization program. The main argument for this limitation is the aspect of "limited time resources". A solution to this problem could therefore be the time-effective and highly individualizable whole-body electromyostimulation (WB-EMS) technology. The aim of the present study is to evaluate the effectiveness of 16 weeks of WB-EMSapplication on maximum strength of the lower extremities, trunk stability and (golf) handicap in male amateur golfers in a (randomized) controlled setting.

ELIGIBILITY:
Inclusion Criteria:

* golf amateurs with a history if golf > 2 years
* no WB-EMS application during the last 12 months

Exclusion Criteria:

* contraindications for WB-EMS (in doubt assessment by study physician)
* contraindications for MRI (in doubt assessment by study physician)
* resistance exercise training for more one 60 min/week during the last 12 months
* expected absence of more than one week during the intervention period (WB-EMS)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
18 hole golf score | through study completion, on average 4 months
  Average golf score of 5 rounds on a 18 hole course (supervised)

SECONDARY OUTCOMES:
Hip-/leg extensor strength | At baseline and after 16 weeks
  Changes of maximum dynamic hip-/leg extensor strength as determine by an isokinetic leg press
Trunk strength | At baseline and after 16 weeks
  Changes of maximum isometric trunk strength (index of trunk extension/-flexion; lateral flexion and trunk rotation) as determined by an isometric testing device
Muscle density at the mid-thigh | At baseline and after 16 weeks
  Muscle density at the mid-thigh as determined by MRI
Muscle density at lumbar spine | At baseline and after 16 weeks
  Muscle density at the para-vertebral site as determined by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Carina Zink-Rückel, MSc, Principal Investigator — Institute of Medical Physics, FAU, Germany
Locations (1):
- Institute of Medical Physics, Friedrich Alexander University Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the responsible researcher [W. Kemmler], upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after publication and ending 3 years following article publication

REFERENCES:
- [Background] Carina Zink-Rückel, Florian Rückel, Simon von Stengel, Wolfgang Kemmler. The Use of Whole Body Electromyostimulation (WB-EMS) as a Golf Warm-Up - A Randomized Controlled Cross-Over Study. Archives of Physical Health and Sports Medicine Volume 2 (2019)1: 04-12